CLINICAL TRIAL: NCT00980421
Title: Effect of Mode of Delivery of Iron and/or Iron and Zinc Supplement on Iron Status Markers and Potential Markers of Iron Toxicity in Children Aged 24-36 Months
Brief Title: Safety of Various Mode of Delivery of Iron Supplement on Iron Toxicity Markers in Preschool Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Annamalai University (Other)
Responsible Party: Dr Venugopal P Menon, Department of Biochemistry and Biotechnology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RHN/NTF/82008-09
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Iron Overload; Oxidative Stress
Keywords: iron; iron toxicity markers; oxidative stress markers; iron supplementation; NTBI; iron over load; interleukin levels; iron status; acut phase reactants; preschool children
MeSH Terms: conditions — Iron Overload | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IT (Experimental): Iron Tablet group (12.5 mg/d) + Placebo Biscuit
  Interventions: Dietary Supplement: Iron Supplementation
- IZ (Experimental): Iron (12.5mg/d)+Zinc (10 mg/d) Tablet Group + Placebo Biscuit
  Interventions: Dietary Supplement: Iron Supplementation
- IB (Experimental): Iron Fortified Biscuit Group(12.5 mg/d)+ Placebo Tablet
  Interventions: Dietary Supplement: Iron Supplementation
- CO (Placebo Comparator): Placebo Tablet + Placebo Biscuit
  Interventions: Dietary Supplement: Iron Supplementation

INTERVENTIONS:
Dietary Supplement: Iron Supplementation — Iron tablet group (12.5 mg/d)+ Placebo Biscuit;Iron(12.5 mg/d)+ Zinc (10 mg/d) tablet group+ Placebo Biscuit; Iron Fortified Biscuit Group (12.5 mg/d)+ Placebo Tablet; Placebo tablet +Placebo Biscuit
  Other Names: Ferrous sulphate

SUMMARY:
The purpose of study is to evaluate and compare the effect of iron supplementation when given as iron tablet or fortified biscuit or combined with zinc in the form of tablet on morbidity and iron toxicity markers among children aged 24-36 months.

DETAILED DESCRIPTION:
The study will be carried out in two phases in Sangam Vihar, Delhi. The survey will be conducted to identify children in the age group of 24-36 months. After obtaining consent, an enrollment form with detailed socio-demographic information about the child will be filled. Blood and urine samples will be collected for estimation of iron status, oxidative stress, immune and interleukin markers. Based on iron status, two randomization lists will be generated i.e. one for iron sufficient and other for iron deficient children. Children will be randomly allocated to receive one of the four interventions (60 in each group) for 180 days. The intervention will be either Iron Tablets (IT) or Iron and Zinc tablets (IZ) or Biscuits fortified with Iron (IB), or Placebo tablets (CO). Children in the iron groups (IT and IB) will receive 12.5 mg/day of iron. Children allocated to receive Iron and Zinc (IZ group) will receive 10 mg/day of Zinc in addition to 12.5 mg/day of Iron. The fortified biscuits (IB) will be formulated by CFTRI, Mysore, India and will have iron in the form of iron sulphate. The iron (IT group) or iron and zinc (IZ group) fortified dispersible tablets will be procured from WHO manufactured by Nutriset (Maluanlay, France). Tablets will have iron salt in the form of ferrous sulphate and zinc in the form of zinc sulphate. The interventions at the baseline on Day 3, on Day 30 (on completion of Phase -I) and on Day 180 (on completion of Phase-II) will be given at the clinic prior to the post 3 hour blood collection. Regular supplementation will be given at home. Children will be followed up on a biweekly basis by the field worker for delivery of the intervention, collection of morbidity and compliance information from the mother/caretaker of the child. During follow-up, blood sample for interleukin levels will be taken in the event of an illness such as diarrhea, pneumonia, fever and severe illness/hospitalization. At the completion of Phase-I (on day 30) and Phase - II (on day 180), the blood and urine samples will be collected again for estimation of iron status, oxidative stress, immune and interleukin markers.

ELIGIBILITY:
Inclusion Criteria:

* between 24-36 months of age
* not severely malnourished or ill requiring hospitalization
* willing to stay in the study area for 6 months
* consent to participate

Exclusion Criteria:

* not consented
* severely malnourished or ill requiring hospitalization

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
The effect of intervention on immune response, iron over load, oxidative stress markers and iron status | 0 month, 1 month and 6 months

SECONDARY OUTCOMES:
Primary Outcome Measures: Mortality Incidence of disease requiring hospitalization interleukin response during severe illness or hospitalization | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Venugopal P Menon, PhD, Principal Investigator — Annamalai University
Locations (1):
- Center for Micronutrient Research, Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Hoppe M, Hulthen L, Hallberg L. The relative bioavailability in humans of elemental iron powders for use in food fortification. Eur J Nutr. 2006 Feb;45(1):37-44. doi: 10.1007/s00394-005-0560-0. Epub 2005 Apr 25. PMID 15864409
- [Background] Olynyk JK, Clarke SL. Iron overload impairs pro-inflammatory cytokine responses by Kupffer cells. J Gastroenterol Hepatol. 2001 Apr;16(4):438-44. doi: 10.1046/j.1440-1746.2001.02456.x. PMID 11354283